CLINICAL TRIAL: NCT05950477
Title: Evaluation of the Association Between Depression and Glycemic Control in People With Type 1 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5733
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2023-06

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Depression Questionnaires — Center of Epidemiological Studies-Depression Scale (CES-D) Patient Health Questionnaire (PHQ-9) Diabetes Treatment Satisfaction Questionnaire (DTSQ) Well-Being Index (WHO-5)

SUMMARY:
Single-center prospective observational pilot study

The aim of the study is to evaluate the potential association between the percentage of time spent in the optimal glycemia range and the score obtained in the questionnaires used to screen for depression.

The study involves only one visit for each participant. Each participant will be asked to sign the informed consent to the study and, during the visit, the following information will be acquired: parameters, history of diabetes, concomitant diseases and medications, and CGM metrics.

The participant will be administered the following questionnaires for the evaluation of depression, patient-reported outcome measure (PROMs) and treatment satisfaction:

* Patient Health Questionnaire (PHQ-9)
* Center of Epidemiological Studies-Depression Scale (CES-D)
* Diabetes Treatment Satisfaction Questionnaire (DTSQ)
* Well-Being Index (WHO-5)
* Problem Areas In Diabetes (PAID-5)
* European Quality of Life, Five Dimension, Five Level (EQ5D5L)

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent before any activity foreseen by the protocol
2. Age > 18 years
3. Subjects with type 1 diabetes mellitus, both on multiple daily injection and with insulin pump, using glucose monitoring systems, both flash glucose monitoring and continuous glucose monitoring

Exclusion criteria:

1. Type 2 diabetes mellitus or other forms of diabetes, such as steroid-induced or secondary to pancreatectomy, pancreatitis, or secondary to endocrinological disorders
2. Previous diagnosis of major depression, bipolar disorder, psychotic disorder, eating disorder (anorexia nervosa, bulimia nervosa, binge eating disorder)
3. Chronic treatment with corticosteroids
4. BMI <19kg/m2
5. Known history of substance or alcohol abuse
6. Patients who have recently been admitted to the psychiatry ward or are being treated with psycho-drugs
7. Conditions that do not allow participation in the activities envisaged by the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 diabetic patients at risk of developing a mood disorders and who meet the inclusion criteria will be enrolled. It is estimated that it is necessary to enroll 100 subjects in order to identify an expected correlation coefficient equal to 0.30, with a power of 85% and a probability value α (two-tailed) of 0.05.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
In 100 subjects with type 1 diabetes it will be evaluated the relationship between time in range, assessed though continuous glucose monitoring, and the score of the depression questionnaire CES-D | 14 days
  Evaluation of the relationship between time in optimal glycemic range (70-180 mg/dl) and scores at depression questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Dario Pitocco, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Università Cattolica del Sacro Cuore, Roma, Italy